CLINICAL TRIAL: NCT02729428
Title: MRI Biomarkers of Risk in Sedentary and Exercise Trained Humans
Brief Title: MRI Biomarkers and Exercise
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2015-1611; CVR-AAA4385 (Other: UW-Madison Study Staff); A176000 (Other: UW, Madison); EDUC/KINESIOLOGY/KINESIO (Other: UW, Madison)
Record Dates: First submitted 2016-03-24; First posted 2016-04-06 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Cerebrovascular Circulation
Keywords: Aging; White Matter Hyperintensity Volume; Default Mode Network Connectivity; Cognitive Function; Cardiorespiratory Fitness; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Exercise trained young adults: Exercise trained young adults between the age of 18-35 years.
  Interventions: Device: MRI
- Sedentary young adults: Sedentary young adults between the age of 18-35 years.
  Interventions: Device: MRI
- Exercise trained older adults: Exercise trained older adults between the age of 55-75 years.
  Interventions: Device: MRI
- Sedentary older adults: Sedentary older adults between the age of 55-75 years.
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — Participants will undergo an MRI scan

SUMMARY:
The overall goal of observational study is to examine the age-related and habitual exercise training status-related differences in structural and functional changes in the human brain, detected by magnetic resonance (MR) imaging.

DETAILED DESCRIPTION:
Normal aging reduces cerebral blood flow, brain volume, and cognitive function, thereby increasing the risk of dementia or Alzheimer's disease. Aging is associated with increased white matter hyperintensities (WMH) and appears to alter functional connectivity within the brain both of which associated with cognitive function (references). Observational studies suggest that regular physical activity is associated with improved cognitive function and higher cerebral blood flow 1,2. However, it is unknown if aging or exercise training status alters the structural and functional biomarkers that are predictive of cognitive decline. Thus, the overall goal of this project is to examine the age-related and exercise training status-related differences in structural and functional changes in the brain, detected by magnetic resonance (MR) imaging.

1. To determine if white matter hyperintensities on MRI scans of the brain are altered by aging and exercise training status.
2. To determine the interaction of aging and habitual physical activity on functional connectivity in the brain.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-35 or 55-75
* Body mass index <34 kg/m2
* Physically active (exercise more than 3 times per week for at least 30 min) or sedentary (no formal exercise over 1 hour per week)

Exclusion Criteria:

* Current smoker
* History or evidence of: hepatic disease, renal disease, hematological disease, peripheral vascular disease, stroke/neurovascular disease, diabetes, hypertension
* Part of a vulnerable population (e.g. pregnant women, prisoner, individuals lacking capacity to consent, etc.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects for this study will include healthy young adults (18-35 years old), sedentary older adults (55-75 years old), and healthy exercise trained older adults (55-75 years old). Both men and women will be eligible to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
White Matter Hyperintensity Volume | 60 minutes
  Utilize an MRI to measure brain volume when participant is at rest

SECONDARY OUTCOMES:
Default Mode Network Connectivity | 60 minutes
  Utilize an MRI to measure functional connectivity in the brain when participant is at rest
Middle Cerebral Artery Blood Flow Scan | 60 minutes
  Utilize an MRI to measure middle cerebral artery blood flow in the brain when the participant is at rest

CONTACTS AND LOCATIONS:
Overall Officials: Jill N Barnes, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Gymnasium-Natatorium, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Erickson KI, Voss MW, Prakash RS, Basak C, Szabo A, Chaddock L, Kim JS, Heo S, Alves H, White SM, Wojcicki TR, Mailey E, Vieira VJ, Martin SA, Pence BD, Woods JA, McAuley E, Kramer AF. Exercise training increases size of hippocampus and improves memory. Proc Natl Acad Sci U S A. 2011 Feb 15;108(7):3017-22. doi: 10.1073/pnas.1015950108. Epub 2011 Jan 31. PMID 21282661
- [Background] Ainslie PN, Cotter JD, George KP, Lucas S, Murrell C, Shave R, Thomas KN, Williams MJ, Atkinson G. Elevation in cerebral blood flow velocity with aerobic fitness throughout healthy human ageing. J Physiol. 2008 Aug 15;586(16):4005-10. doi: 10.1113/jphysiol.2008.158279. Epub 2008 Jul 17. PMID 18635643
- [Background] Bakker SL, de Leeuw FE, den Heijer T, Koudstaal PJ, Hofman A, Breteler MM. Cerebral haemodynamics in the elderly: the rotterdam study. Neuroepidemiology. 2004 Jul-Aug;23(4):178-84. doi: 10.1159/000078503. PMID 15272220
- [Background] Selim M, Jones R, Novak P, Zhao P, Novak V. The effects of body mass index on cerebral blood flow velocity. Clin Auton Res. 2008 Dec;18(6):331-8. doi: 10.1007/s10286-008-0490-z. Epub 2008 Aug 22. PMID 18726054
- [Background] Dandona P, James IM, Newbury PA, Woollard ML, Beckett AG. Cerebral blood flow in diabetes mellitus: evidence of abnormal cerebrovascular reactivity. Br Med J. 1978 Jul 29;2(6133):325-6. doi: 10.1136/bmj.2.6133.325. PMID 687900
- [Background] Barnes JN, Schmidt JE, Nicholson WT, Joyner MJ. Cyclooxygenase inhibition abolishes age-related differences in cerebral vasodilator responses to hypercapnia. J Appl Physiol (1985). 2012 Jun;112(11):1884-90. doi: 10.1152/japplphysiol.01270.2011. Epub 2012 Mar 22. PMID 22442028
- [Background] Lipsitz LA, Mukai S, Hamner J, Gagnon M, Babikian V. Dynamic regulation of middle cerebral artery blood flow velocity in aging and hypertension. Stroke. 2000 Aug;31(8):1897-903. doi: 10.1161/01.str.31.8.1897. PMID 10926954
- [Background] Kearney-Schwartz A, Rossignol P, Bracard S, Felblinger J, Fay R, Boivin JM, Lecompte T, Lacolley P, Benetos A, Zannad F. Vascular structure and function is correlated to cognitive performance and white matter hyperintensities in older hypertensive patients with subjective memory complaints. Stroke. 2009 Apr;40(4):1229-36. doi: 10.1161/STROKEAHA.108.532853. Epub 2009 Feb 26. PMID 19246701
- [Background] Smith EE, Greenberg SM. Beta-amyloid, blood vessels, and brain function. Stroke. 2009 Jul;40(7):2601-6. doi: 10.1161/STROKEAHA.108.536839. Epub 2009 May 14. PMID 19443808
- [Background] Barnes JN, Taylor JL, Kluck BN, Johnson CP, Joyner MJ. Cerebrovascular reactivity is associated with maximal aerobic capacity in healthy older adults. J Appl Physiol (1985). 2013 May 15;114(10):1383-7. doi: 10.1152/japplphysiol.01258.2012. Epub 2013 Mar 7. PMID 23471946
- [Background] Girouard H, Iadecola C. Neurovascular coupling in the normal brain and in hypertension, stroke, and Alzheimer disease. J Appl Physiol (1985). 2006 Jan;100(1):328-35. doi: 10.1152/japplphysiol.00966.2005. PMID 16357086
- [Background] Geda YE, Roberts RO, Knopman DS, Christianson TJ, Pankratz VS, Ivnik RJ, Boeve BF, Tangalos EG, Petersen RC, Rocca WA. Physical exercise, aging, and mild cognitive impairment: a population-based study. Arch Neurol. 2010 Jan;67(1):80-6. doi: 10.1001/archneurol.2009.297. PMID 20065133
- [Background] Baker LD, Frank LL, Foster-Schubert K, Green PS, Wilkinson CW, McTiernan A, Cholerton BA, Plymate SR, Fishel MA, Watson GS, Duncan GE, Mehta PD, Craft S. Aerobic exercise improves cognition for older adults with glucose intolerance, a risk factor for Alzheimer's disease. J Alzheimers Dis. 2010;22(2):569-79. doi: 10.3233/JAD-2010-100768. PMID 20847403
- [Background] Lautenschlager NT, Cox KL, Flicker L, Foster JK, van Bockxmeer FM, Xiao J, Greenop KR, Almeida OP. Effect of physical activity on cognitive function in older adults at risk for Alzheimer disease: a randomized trial. JAMA. 2008 Sep 3;300(9):1027-37. doi: 10.1001/jama.300.9.1027. PMID 18768414
- [Background] Galetta F, Franzoni F, Plantinga Y, Ghiadoni L, Rossi M, Prattichizzo F, Carpi A, Taddei S, Santoro G. Ambulatory blood pressure monitoring and endothelium-dependent vasodilation in the elderly athletes. Biomed Pharmacother. 2006 Sep;60(8):443-7. doi: 10.1016/j.biopha.2006.07.013. Epub 2006 Aug 2. PMID 16904861
- [Background] Franzoni F, Ghiadoni L, Galetta F, Plantinga Y, Lubrano V, Huang Y, Salvetti G, Regoli F, Taddei S, Santoro G, Salvetti A. Physical activity, plasma antioxidant capacity, and endothelium-dependent vasodilation in young and older men. Am J Hypertens. 2005 Apr;18(4 Pt 1):510-6. doi: 10.1016/j.amjhyper.2004.11.006. PMID 15831361
- [Background] Green DJ, O'Driscoll G, Joyner MJ, Cable NT. Exercise and cardiovascular risk reduction: time to update the rationale for exercise? J Appl Physiol (1985). 2008 Aug;105(2):766-8. doi: 10.1152/japplphysiol.01028.2007. Epub 2008 Jan 3. No abstract available. PMID 18174390
- [Background] Seifert T, Brassard P, Wissenberg M, Rasmussen P, Nordby P, Stallknecht B, Adser H, Jakobsen AH, Pilegaard H, Nielsen HB, Secher NH. Endurance training enhances BDNF release from the human brain. Am J Physiol Regul Integr Comp Physiol. 2010 Feb;298(2):R372-7. doi: 10.1152/ajpregu.00525.2009. Epub 2009 Nov 18. PMID 19923361
- [Background] van Dijk EJ, Prins ND, Vrooman HA, Hofman A, Koudstaal PJ, Breteler MM. Progression of cerebral small vessel disease in relation to risk factors and cognitive consequences: Rotterdam Scan study. Stroke. 2008 Oct;39(10):2712-9. doi: 10.1161/STROKEAHA.107.513176. Epub 2008 Jul 17. PMID 18635849
- [Background] Raz N, Yang Y, Dahle CL, Land S. Volume of white matter hyperintensities in healthy adults: contribution of age, vascular risk factors, and inflammation-related genetic variants. Biochim Biophys Acta. 2012 Mar;1822(3):361-9. doi: 10.1016/j.bbadis.2011.08.007. Epub 2011 Aug 25. PMID 21889590
- [Background] Kantarci K, Weigand SD, Przybelski SA, Shiung MM, Whitwell JL, Negash S, Knopman DS, Boeve BF, O'Brien PC, Petersen RC, Jack CR Jr. Risk of dementia in MCI: combined effect of cerebrovascular disease, volumetric MRI, and 1H MRS. Neurology. 2009 Apr 28;72(17):1519-25. doi: 10.1212/WNL.0b013e3181a2e864. PMID 19398707
- [Background] Silbert LC, Nelson C, Howieson DB, Moore MM, Kaye JA. Impact of white matter hyperintensity volume progression on rate of cognitive and motor decline. Neurology. 2008 Jul 8;71(2):108-13. doi: 10.1212/01.wnl.0000316799.86917.37. PMID 18606964
- [Background] Rosano C, Watson N, Chang Y, Newman AB, Aizenstein HJ, Du Y, Venkatraman V, Harris TB, Barinas-Mitchell E, Sutton-Tyrrell K. Aortic pulse wave velocity predicts focal white matter hyperintensities in a biracial cohort of older adults. Hypertension. 2013 Jan;61(1):160-5. doi: 10.1161/HYPERTENSIONAHA.112.198069. Epub 2012 Nov 19. PMID 23172923
- [Background] Raichle ME, MacLeod AM, Snyder AZ, Powers WJ, Gusnard DA, Shulman GL. A default mode of brain function. Proc Natl Acad Sci U S A. 2001 Jan 16;98(2):676-82. doi: 10.1073/pnas.98.2.676. PMID 11209064
- [Background] Greicius MD, Krasnow B, Reiss AL, Menon V. Functional connectivity in the resting brain: a network analysis of the default mode hypothesis. Proc Natl Acad Sci U S A. 2003 Jan 7;100(1):253-8. doi: 10.1073/pnas.0135058100. Epub 2002 Dec 27. PMID 12506194
- [Background] Chen G, Ward BD, Xie C, Li W, Wu Z, Jones JL, Franczak M, Antuono P, Li SJ. Classification of Alzheimer disease, mild cognitive impairment, and normal cognitive status with large-scale network analysis based on resting-state functional MR imaging. Radiology. 2011 Apr;259(1):213-21. doi: 10.1148/radiol.10100734. Epub 2011 Jan 19. PMID 21248238
- [Background] Jones DT, Machulda MM, Vemuri P, McDade EM, Zeng G, Senjem ML, Gunter JL, Przybelski SA, Avula RT, Knopman DS, Boeve BF, Petersen RC, Jack CR Jr. Age-related changes in the default mode network are more advanced in Alzheimer disease. Neurology. 2011 Oct 18;77(16):1524-31. doi: 10.1212/WNL.0b013e318233b33d. Epub 2011 Oct 5. PMID 21975202
- [Background] Andrews-Hanna JR, Snyder AZ, Vincent JL, Lustig C, Head D, Raichle ME, Buckner RL. Disruption of large-scale brain systems in advanced aging. Neuron. 2007 Dec 6;56(5):924-35. doi: 10.1016/j.neuron.2007.10.038. PMID 18054866
- [Background] Damoiseaux JS, Beckmann CF, Arigita EJ, Barkhof F, Scheltens P, Stam CJ, Smith SM, Rombouts SA. Reduced resting-state brain activity in the "default network" in normal aging. Cereb Cortex. 2008 Aug;18(8):1856-64. doi: 10.1093/cercor/bhm207. Epub 2007 Dec 5. PMID 18063564
- [Background] Voss MW, Erickson KI, Prakash RS, Chaddock L, Malkowski E, Alves H, Kim JS, Morris KS, White SM, Wojcicki TR, Hu L, Szabo A, Klamm E, McAuley E, Kramer AF. Functional connectivity: a source of variance in the association between cardiorespiratory fitness and cognition? Neuropsychologia. 2010 Apr;48(5):1394-406. doi: 10.1016/j.neuropsychologia.2010.01.005. Epub 2010 Jan 15. PMID 20079755